CLINICAL TRIAL: NCT07074821
Title: Effect of Tunneled Hemodialysis Catheter Antimicrobial Lock Solution in Prevention of Catheter Related Blood Stream Infection.
Brief Title: Antimicrobial Locks for Hemodialysis Catheter Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oman Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Ahmed Said Mohammed, Principal investigator, Oman Ministry of Health
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MoH/CSR/24/27480
Record Dates: First submitted 2025-05-04; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Catheter Related Blood Stream Infection; Hemodialysis; Vascular Access
Keywords: catheter related infection; hemodialysis; Taurolidine
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) patients used usual Heparin used as tunneled hemodialysis lock solution (No Intervention): Measure incidence of catheter related blood stream infection while patients use Heparin as catheter lock
- Group (B) patients used Taurolidine based lock solution as tunneled hemodialysis catheter lock (Experimental): Measure incidence of catheter related blood stream infection while patients use Taurolidine based lock solution as catheter lock
  Interventions: Drug: Taurolidine citrate 4% and heparin 500

INTERVENTIONS:
Drug: Taurolidine citrate 4% and heparin 500 — Taurolidine ,citrate 4% and heparin 500 units per ml used as lock solution in tunneled hemodialysis catheter
  Arms: Group (B) patients used Taurolidine based lock solution as tunneled hemodialysis catheter lock

SUMMARY:
Tunneled hemodialysis catheters are susceptible to infection with high incidence of complication to the hemodialysis patients .The study aimed to prevent catheter infection through comparing use of antimicrobial solution (Taurolidine) when used as lock solution installed in the lumen of the catheter at the end of the hemodialysis session with the usually used lock solution heparin. The Study was performed on 100 hemodialysis patients over one year in Sohar hospital ,Oman .

ELIGIBILITY:
Inclusion criteria:

- All clinically stable adult end stage renal disease patients commence regular hemodialysis through tunneled hemodialysis catheter at Sohar hospital hemodialysis unit.

Exclusion criteria:

* Patients with difficult vascular access and the tunneled hemodialysis catheter is the only functioning vascular access .
* Patients with poor flow from the catheter.
* Patients with active infection .
* Patients have displayed allergic reactions to either citrate or taurolidine.
* Patients were taking medication incompatible with either citrate or taurolidine

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Comparison between both groups in terms of incidence of Catheter related blood stream infection | one year
  The investigators have studied the incidence of catheter related bacterial infection in both groups to determine superior effectiveness of Taurolidine lock solution than Heparin lock only in terms of prevention of infection .

SECONDARY OUTCOMES:
Comparison between both groups in terms of treatment cost | one year
  The secondary outcome measure was to compare the treatment cost in both groups to determine cost effectiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Sohar hospital, Sohar, Sohar, Oman

IPD SHARING:
Plan to Share IPD: Yes
Methodology and results